CLINICAL TRIAL: NCT02724631
Title: Evaluation of Efficacy of Use of TubeClear® to Restore Patency to Occluded Enteral Access Devices in Pediatric Patients (Phase I)
Brief Title: TubeClear® Evaluation in Pediatric Patients (Phase I)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit; study determined not feasible to continue
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Actuated Medical, Inc. (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-011488; 5R44HD065365-04 (NIH)
Record Dates: First submitted 2016-03-14; First posted 2016-03-31 (Estimated); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Enteral Nutrition
Keywords: Clogged enteral access devices; Occluded enteral access device; Enteral nutrition; Enteral access device; Tube Feeding; Gastric Feeding Tubes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TubeClear® (Phase I) (Experimental): To determine feasibility and tolerability, 15 subjects will receive the TubeClear® intervention. If the TubeClear® intervention is unable to restore Enteral Access Device patency, further steps to restore patency of the occluded EAD will be determined by the clinical team per usual practice.
  Interventions: Device: TubeClear® intervention

INTERVENTIONS:
Device: TubeClear® intervention — The TubeClear® device is deemed by the Food and Drug Administration (FDA) to be non-significant risk (NSR) for use in this study. It is a control box and a single use clearing stem used to resolve the clog in an enteral access device within five minutes following the intervention.

SUMMARY:
This is the first of three planned phases designed to evaluate the feasibility and tolerability of TubeClear® to restore patency in occluded Pediatric Enteral Access Devices. Based on preliminary data obtained from this phase of the study, subsequent phases will continue to evaluate feasibility and tolerability (Phase IIA) and ultimately compare efficacy of TubeClear® to the Children's Hospital of Philadelphia (CHOP) Standard Treatment to restore patency in occluded Pediatric Enteral Access Devices (EAD) (Phase IIB).

DETAILED DESCRIPTION:
Occluded enteral access devices (EADs) are a significant problem for pediatric patients, with occlusion rates ranging from 12.5% to 35%. Occluded EADs can lead to extended times of decreased energy intake, resulting in patients quickly exhausting their energy reserves and developing dehydration with electrolyte abnormalities. Current methods used to restore patency to an occluded EAD at The Children's Hospital of Philadelphia (CHOP) involve application of enzymes and chemicals (e.g., Clog Zapper), which have variable rates of timely success. If these methods are unsuccessful and patency cannot be restored, the EAD must be replaced and may require radiological intervention with exposure to radiation and contrast material. TubeClear® addresses this clinical need to safely and efficaciously restore patency to occluded EADs at the patients' bedside while the EAD remains in the patient. Additionally, this reduces the need to transport the patient to the radiology suite with subsequent exposure to radiation and contrast material for EAD location conformation after replacement.

Current Study (Phase I): Feasibility and tolerability of TubeClear® intervention in 15 consecutive eligible Subjects with occluded Enteral Access Devices who have not attained their 18th birthday.

Following successful completion of Phase I as deemed by the Institutional Review Board (IRB), the Study will proceed to Phase IIA and IIB to run concurrently.

Future Studies:

Phase IIA: Ability of TubeClear® intervention to restore patency in 15 consecutive eligible Subjects with occluded Enteral Access Devices who have not attained their 11th birthday.

Phase IIB: Randomized efficacy comparison between 17 subjects using the TubeClear® intervention and 17 subjects using CHOP Standard Treatment in eligible Subjects with occluded Enteral Access Devices who are between 11 years of age and have not attained their 18th birthday.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between who have not attained their 18th birthday
2. Indwelling occluded EAD(P) that is either:

   * Nasoduodenal Tube (ND), Nasogastric Tube (NG), Nasojejunal Tube (NJ) composed of Polyvinyl Chloride (PVC) and Polyurethane 6 - 8 Fr, 38 - 140 cm cm; or
   * Nasogastric Tube (NG) (Corflo, Corpak MedSystems) used as a jejunal tube inserted through a gastrostomy tube, 6 - 8 Fr, 38 - 140 cm
   * GJ (AMT) 14 Fr, 38 - 140 cm (15 - 55 in)

Exclusion Criteria:

1. Ward of the state
2. Positive pregnancy test/ Pregnant females
3. Any active gastrointestinal abnormalities or malformations, including but not limited to infections, inflammation, obstruction and/or recent abdominal surgery or trauma
4. Constant dependency on the EAD(P) for a glucose source (e.g. hyperinsulinism states)
5. Unable to tolerate water volume needed for the EAD(P) flush
6. Allergies to the contrast agent(s) used in post-Intervention radiological imaging
7. Measured total length of EAD(P) less than 38 cm (15 inches) - from external port to EAD(P) distal end
8. Unknown length of EAD(P)
9. Attending physician declines enrollment based on clinical judgement
10. Subject attains 18 years of age during study duration

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Srinivasan, MBBS, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are pediatric patients (Less than age 18) and are admitted to the Children's Hospital of Philadelphia (CHOP) Pediatric Intensive Care Unit (PICU), Progressive Care Unit (PCU), or Interventional Radiology (IR) with an existing or a newly inserted Pediatric Enteral Access Device (EAD(P)) that becomes occluded. Occlusion is defined by direct identification of a clog or through a feeding pump alarm that sounds when patency of an EAD(P) is disrupted.
Pre-assignment Details: Only 1 participant was enrolled. Unable to restore patency to indwelling feeding device. The study was terminated due to lack of enrollment; insufficient data for analysis to assess outcome or draw conclusions from the intervention.
Period: Overall Study
Arm/Group | TubeClear® (Phase I)
Started | 1
Completed | 0
Not Completed | 1
Not completed — unable to clear indwelling feeding tube device | 1

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled. Unable to restore patency to indwelling feeding device. The study was terminated due to lack of enrollment; insufficient data for analysis to assess outcome or draw conclusions from the intervention
Arm/Group | TubeClear® (Phase I)
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years of age | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Successful Attempts to Restore EAD(P) Patency
Description: Feasibility will be defined as ability of the user to operate TubeClear® from clearing stem insertion into the occluded Enteral Access Device through activation to patency restoration. Successful restoration of patency will be defined as the ability to flush the EAD(P) with 10ml of air within five minutes following the intervention by the investigator.
Time Frame: Baseline to 5 minutes post-intervention
Population: as for baseline characteristics
Arm/Group | TubeClear® (Phase I)
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Age-Appropriate Pain Score
Description: Tolerability will be defined as ability of the subject to undergo TubeClear® intervention. To assess this, subject pain will be assessed before and after use of TubeClear® intervention and then daily for up to 3 days post-intervention using one of the well-established age-appropriate pain scales. Based on subject age, one of the following pain scale assessments will be used: Face, Legs, Activity, Cry, Consolability (FLACC) Scale; Revised Face, Legs, Activity, Cry, Consolability (rFLACC) scale; FACES pain scale revised (FPS-R); Numeric Pain Scale; or Nursing Judgement
Time Frame: Baseline to 3 days post-intervention
Population: as for baseline characteristics
Arm/Group | TubeClear® (Phase I)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Time frame = 5 minutes
Arm/Group | TubeClear® (Phase I)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study ended due to inability to recruit applicable subjects to trial the study intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT02724631/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT02724631/ICF_001.pdf